CLINICAL TRIAL: NCT05997849
Title: Development of a Multiplatform Mobile Tool for the Prevention of Mental Health Pathologies in Chilean Adults
Brief Title: Development of a Multiplatform Mental Health Mobile Tool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Talca (Other)
Collaborators: Gobierno Regional del Maule (Unknown)
Responsible Party: Principal Investigator, Nadia Ramos Álvarado, Assistant Professor, University of Talca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FIC 40027682
Record Dates: First submitted 2023-08-04; First posted 2023-08-18 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Depression; Anxiety
Keywords: Mental health; Mobile application; Depression; Anxiety; RCT
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The study uses a parallel model for the delivery of the interventions, where the application-based interventions will be carried out simultaneously for all groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: Masking of the participants will be achieved by assigning them to intervention groups without stating the content or purpose of said group beyond the general guidelines of knowing that the intervention is mental health related. Masking of the outcome assessors will be achieved by providing them an Anonymized participant database after the application period and recollection of data has ended.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Monitoring and psychoeducation module (Active Comparator): The participants in this group will have access only to the monitoring and psychoeducation module for 30 days. The monitoring module consists of a set of self-report measures, and the psychoeducation is delivered through videos.
  Interventions: Behavioral: Mobile application
- Mindfulness strategies module (Experimental): Participants in this group will have access to the monitoring, psychoeducation and mindfulness strategies modules for 30 days. The mindfulness strategies module includes a set of mindfulness-based self-guided techniques for depression and anxiety symptoms. These techniques are delivered in three steps: Learning, Understanding and Practicing.
  Interventions: Behavioral: Mobile application
- Behavioral activation strategies module (Experimental): Participants in this group will have access to the monitoring, psychoeducation and mindfulness strategies modules for 30 days. The behavioral activation strategies module includes a set of behavioral activation self-guided techniques for depression and anxiety symptoms. These techniques are delivered in three steps: Learning, Understanding and Practicing.
  Interventions: Behavioral: Mobile application
- Cognitive strategies module (Experimental): Participants in this group will have access to the monitoring, psychoeducation and mindfulness strategies modules for 30 days. The mindfulness strategies module includes a set of cognitive-based self-guided techniques for depression and anxiety symptoms, derived from CBT guidelines. These techniques are delivered in three steps: Learning, Understanding and Practicing.
  Interventions: Behavioral: Mobile application

INTERVENTIONS:
Behavioral: Mobile application — A mobile application for the management of anxiety and depressive symptoms through self-applied emotional regulation tools.

SUMMARY:
Mobile applications for mental health (MAMH) have shown great potential for delivering digital interventions for the general population. However, most of these apps do not have evidence on how they work. Thus, users may be exposed to products that do not offer any real benefit, or that could harm them.

Similarly, the most popular MAMHs use several techniques to deliver their mental health content, but it is still necessary to identify how effective each component is, so that these interventions can be optimized.

The aim of this clinical trial is to evaluate how effective the components of evaluation, psychoeducation, and emotional regulation strategies are in a multiplatform MAMH in Chile. 196 adults will have access to different components of the application after consenting to participate in the study. They will be randomly assigned to one of four groups and will use the mobile app for a fixed period. Researchers will compare depressive and anxiety symptoms between the adults in these groups, will either receive:

1. Psychoeducation.
2. Psychoeducation and mindfulness strategies.
3. Psychoeducation and behavioral activation strategies.
4. Psychoeducation and cognitive strategies.

All groups will be continuously assessed and monitored. The researchers hypothesize that the psychoeducation combined with any set of self-regulatory strategies will prove more effective than the psychoeducation component alone in decreasing symptomatology.

DETAILED DESCRIPTION:
Anxiety and depressive symptoms are prevalent in Chilean adults. The considerable gaps in health-related demand and medical-care supply hinders the access to psychological treatment, which negatively impacts the population's overall well-being. In this scenario, it becomes necessary to find alternatives that enable the access to mental health treatment. The use of remote psychological treatments, particularly mobile applications for mental health (MAMH), has been deemed as promising in this regard. Although in recent years the number of MAMH has increased explosively, many of them do not have any theoretical support for their effectiveness. The few MAHMs that have presented evidence of their effectiveness reducing symptomathology use the elements of assessment, psychoeducation, and symptom-management strategies as intervention pillars. The combination of these three elements seems to be highly effective, but no studies have examined the effectiveness of said components in detail. Thus, the aim of this exploratory study is to develop a multiplatform mobile application for mental health care for adults, and test the effectiveness of its assessment, psychoeducation, and emotional regulation strategy components, at post-intervention and 1-month follow-up. In the study, 4 experimental conditions are carried out to evaluate the components both in their effectiveness, and their usability and applicability. The researchers hypothesize that the combination of psychoeducation and any self-regulatory strategies will prove more effective than the evaluation and psychoeducation component alone in decreasing symptomatology.

The expected sample comprises a total 196 participants equally divided in the 4 groups, that will actively test the application. In Group 1: the participants will have access only to the monitoring (or evaluation) and psychoeducation module for 30 days; Group 2: participants will have access to the monitoring module, psychoeducation and mindfulness strategies for 30 days; Group 3: participants will have access to the monitoring module, psychoeducation and behavioral activation strategies for 30 days; Group 4: Participants will have access to the monitoring, psychoeducation and cognitive strategies module for 30 days. Outcomes measured will consider self-reported anxiety and depressive symptoms, among other psychological and well-being variables. These outcomes will be measured at pre-intervention, post-intervention, and 1-month follow-up. Participants will be randomly assigned to any group with a 1:1 allocation as per computer-generated randomization, using the PHP rand() function. Additionally, a subsample of 32 random participants will also engage in focus-groups to assess user experience with the application. Analyses of all outcomes at different timepoints will be carried out through linear mixed model for repeated measures (MMRM) analyses, and content analyses. This study is expected to last 14 months (September 2023 to October 2024).

ELIGIBILITY:
Inclusion Criteria:

* Adult Chilean citizens, 18 years old or older.
* With access to a computer, tablet, or smartphone (Android or iOS) with Internet.
* No diagnosed mental health problems or
* With a diagnosed mental health problem undergoing treatment. The mental health diagnosis and current treatment will be assessed solely by the participant's self-report.

Exclusion Criteria:

* Individuals with substance abuse problems, psychotic symptoms, organic brain disorders (e.g., dementia), self-harm or harm to others, or serious health problems that prevent the use of the application.
* Participants reporting scores greater than 1 on question 9 (suicidal ideation) on the PHQ-9

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2025-01-24 (Actual)

PRIMARY OUTCOMES:
Anxiety symptoms | Measured at baseline (pre-intervention), immediately after the intervention, and at 1-month follow-up for all groups. Monitoring of anxiety symptoms is carried out with PHQ-4 on a weekly basis.
  Current anxiety symptoms as measured by Generalized Anxiety Disorder Scale - 7 (Generalized Anxiety Disorder-7). It consists of 7 items that the person assesses on a scale of 0 to 3 according to the frequency with which each symptom has disturbed them during the last 2 weeks (Spitzer et al., 2006). (2) The PHQ-4 instrument (Kroenke, Spitzer, Williams & Löwe, 2009) has 4 items that assess depressive and anxiety symptoms in the last week.
Depressive symptoms | Measured at baseline (pre-intervention), immediately after the intervention, and at 1-month follow-up for all groups. Monitoring of depressive symptoms is carried out with PHQ-4 on a weekly basis.
  Current depressive symptoms as measured by PHQ-9 depression scale (Patient Health Questionnaire) consists of 9 items that evaluate the presence of depressive symptoms present in the last 2 weeks; with a response scale of 0 ="never", 1 = "some days", 2 = "more than half the days" and 3 = "almost every day". It presents a Cronbach's alpha of 0.83 in the Chilean sample (Baader et al., 2012). (2) The PHQ-4 instrument (Kroenke, Spitzer, Williams & Löwe, 2009) has 4 items that assess depressive and anxiety symptoms in the last week.

SECONDARY OUTCOMES:
Wellbeing | Measured at baseline (pre-intervention), immediately after the intervention, and at 1-month follow-up for all groups.
  Perceived psychological and overall wellbeing is measured by PHI Scale (Pemberton Happiness Index): 21-item instrument, evaluates in 2 subscales, psychological well-being (experienced, 5 positive experiences and 5 negative experiences) and subjective well-being (remembered). The scale is Likert-type, with scores per item from 0 to 10 (Paiva et al., 2016).
Resilience | Measured at baseline (pre-intervention), immediately after the intervention, and at 1-month follow-up for all groups.
  Perceived resilience as measured by the BRS (Brief Resilience Scale), a 6-item instrument, Likert score from 1 to 5. It has three inverted items and the rating results from the average of the scores obtained (Smith et al., 2008).
Ruminative thoughts | Measured at baseline (pre-intervention), immediately after the intervention, and at 1-month follow-up for all groups.
  Rumination and ruminative thoughts are assessed by the Ruminative Response Scale (RRS Short version), consisting of 10 items that measure ruminant thoughts in two dimensions: reflection and restlessness. It has a high level of internal consistency (Cronbach's a = .85). Each item is scored on a 4-point Likert scale from 1 (almost never) to 4 (almost always) (Treynor, Gonzalez & Nolen-Hoeksema, 2003).
Emotion regulation | Measured at baseline (pre-intervention), immediately after the intervention, and at 1-month follow-up for all groups.
  Emotion regulation is assessed by the Emotional Regulation Questionnaire (ERQ), a 10-item questionnaire designed to measure respondents' tendency to regulate their emotions in two ways: (1) Cognitive Reappraisal (1,3,5,7,8,10) and (2) Expressive suppression (2, 4, 6, 9) (Gross & John, 2003).
Mindfulness skills | Measured at baseline (pre-intervention), immediately after the intervention, and at 1-month follow-up for all groups.
  Assessed with MAAS (Mindfulness attention awareness scale), an instrument composed of 14 items, Likert score from 1 to 6. The scores obtained are added and the higher the score, the greater the ability to pay attention fully and consciously. The average scores of the non-clinical participants tend to be around 65 points out of a total of 84. (Brown & Ryan, 2003)

CONTACTS AND LOCATIONS:
Overall Officials: Nadia A Ramos, PhD, Principal Investigator — University of Talca
Locations (1):
- Universidad de Talca, Talca, Maule Region, Chile

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD and any supporting information will be made available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD and any supporting information will be available starting 6 months after publication of study results.
Access Criteria: Any researcher can contact the lead investigator (NR) and request access for all raw data.

REFERENCES:
- [Background] Torous, J., Levin, M. E., Ahern, D. K., & Oser, M. L. (2017). Cognitive Behavioral Mobile Applications: Clinical Studies, Marketplace Overview, and Research Agenda. Cognitive and Behavioral Practice, 24(2), 215-225. https://doi.org/10.1016/j.cbpra.2016.05.007
- [Background] Stawarz K, Preist C, Tallon D, Wiles N, Coyle D. User Experience of Cognitive Behavioral Therapy Apps for Depression: An Analysis of App Functionality and User Reviews. J Med Internet Res. 2018 Jun 6;20(6):e10120. doi: 10.2196/10120. PMID 29875087
- [Background] Lagan S, D'Mello R, Vaidyam A, Bilden R, Torous J. Assessing mental health apps marketplaces with objective metrics from 29,190 data points from 278 apps. Acta Psychiatr Scand. 2021 Aug;144(2):201-210. doi: 10.1111/acps.13306. Epub 2021 Apr 29. PMID 33835483